CLINICAL TRIAL: NCT02413307
Title: The Development and Evaluation of a Brief Self-practice Compassion Focused Therapy (CFT) Intervention as an Adjunct to TAU for Trauma Patients
Brief Title: The Development and Evaluation of a Brief CFT Intervention for Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lincoln (Other)
Collaborators: University of Nottingham (Other)
Responsible Party: Principal Investigator, Claire Rycroft, Clinical Psychologist, University of Lincoln
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 160094
Record Dates: First submitted 2015-04-06; First posted 2015-04-09 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Trauma; PTSD
Keywords: Compassion Focused Therapy
MeSH Terms: conditions — Wounds and Injuries; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): Self-practice compassion focused therapy intervention following written or audio scripts. This includes instructions, an explanation of compassion and aims of the intervention. It includes several exercises designed to increase self-compassion including breathing exercises and compassionate imagery exercises focused on self and others
  Interventions: Other: Compassion Focused Therapy (self-practice)
- Waiting List Control (No Intervention): Participants on the waiting list for trauma specific therapy. These will be participants who have consented to engaging in the research project but their intervention phase has a delayed start.

INTERVENTIONS:
Other: Compassion Focused Therapy (self-practice) — Daily practice of the CFT exercises for a minimum of five minutes per day. This is completed for a period of three weeks.
  Arms: Intervention Group

SUMMARY:
**PLEASE NOTE** this study is currently open only to clients on the waiting list at the Centre for Trauma Resilience and Growth, UK.

The project will involve adapting and implementing a five minute daily self-practice compassion-focused intervention and evaluate its impact on psychological and physiological factors associated with trauma. It aims to offer a novel intervention which may facilitate further benefits from trauma specific therapy. This would be a unique use of self-practice Compassion Focused Therapy (CFT) specifically for trauma clients. Previous research has found that many factors can impact on client's benefitting from therapy, including depression, anxiety and self-criticism. These things also get in the way of being compassionate towards oneself, and this can be a difficulty for people who have experienced traumatic events. Service users have identified that additional support before trauma specific therapy can be useful and this may offer a positive use of time whilst on therapy waiting lists.

Hypotheses:

i. A brief CFT intervention will decrease levels of depression, anxiety, stress and increase baseline Heart Rate Variability.

ii. The compassion focused intervention will increase experiences of self-compassion, social safeness, and reduce levels of self-criticism.

iii. High 'fear of compassion' will moderate the impact of the intervention and result in smaller changes in depression, anxiety, stress and post traumatic change.

Clients of the Centre for trauma, resilience and growth will be approached to participate in the study. All participants will have experienced trauma for which they are seeking psychological support. The current compassion focused intervention will be offered to participants on the waiting list for trauma specific therapy at the trauma centre. Each participant will be asked to practice the intervention in their own time over a period of three weeks. There will be initial assessments, repeated assessments following the intervention, and repeated assessments pre and post trauma specific therapies engaged in.

DETAILED DESCRIPTION:
The project will implement a five-minute daily self-practice CFT intervention and evaluate its impact on psychological and physiological factors associated with trauma. It aims to offer a novel intervention which may facilitate further benefits from trauma-specific therapy. Follow-up data may demonstrate maintenance of positive effects and increased positive effects if self-practice is continued. This would be a unique use of self-practice CFT specifically for trauma clients.

Study Design The study will use a delayed intervention Randomised Controlled Trial (RCT) using a block design.A delayed intervention group will act as a passive control group. Participants will engage in a daily five-minute self-practice CFT intervention prior to engaging in trauma-specific TAU. The CFT intervention will be adapted specifically for trauma clients based on the literature review, involvement of service users, and close collaboration with Professor Paul Gilbert. The project will involve three stages, outlined below.

Stage One: Development of CFT intervention and feasibility testing

Development The final version of the adapted five-minute CFT practice will include consultation with Paul Gilbert as original author of the five-minute CFT intervention (unpublished) as well as consultation with research supervisors. It will be available in both audio and written format. Permission has kindly been given by Paul Gilbert to adapt this for use in the project.

The current version of the CFT intervention includes: instructions, an explanation of compassion and aims of the intervention. It includes several exercises designed to increase self-compassion including breathing exercises and compassionate imagery exercises focused on self and others.

Throughout the adaptation process, services users' ideas will be considered. The intervention will include explicit instructions not to focus on traumatic events participants have experienced. This will be addressed in their trauma-specific therapy . Participants will be encouraged to focus on milder difficulties and stressors. The adaptations will account for the current literature in CFT and maintain its basic principles, focusing on building self-compassion and reducing self-criticism.

Participant sampling for feasibility testing will be opportunistic, seeking voluntary engagement from clients currently accessing services. The sample size for this stage is not explicitly defined and will depend on the number of interested parties. This aims to test feasibility and acceptability of the intervention and its instructions with a clinical population. Participants will be asked to practice the intervention over a two-week period.

Stage Two: Randomised controlled trial Design The research will utilise a single-blind blocked-randomisation design, incorporating three-week intervention versus waiting-list blocks. Following the end of the initial block, participants who formed the passive, waiting-list group will engage in the active intervention, whilst the active group will continue to remain on the waiting list. Both routine and project-specific outcomes measures will be implemented.

Therapists from the recruitment site will conduct screening assessments and post TAU assessments. All other measurements will be completed with the primary researcher. Prospective participants will be provided with an information sheet as part of the screening interview and, if they consent, will be contacted by the researcher. They will be given the opportunity to ask questions and be asked to sign a consent form if they wish to participate. It will be made clear that non-participation will have no adverse effects on their access to psychological treatment and that engaging in the project will not affect their access to treatment. An initial appointment will then be made and the pre-intervention assessments completed. Participants will be allocated to the CFT or waiting-list condition using blocked randomisation. Self-report measures will be uploaded to an academically-focused online survey tool (eSurv) and participants will have Heart Rate Variability (HRV) measurements taken during face-to-face appointments with the primary researcher.

The five-minute CFT self-practice intervention will be available both in written and audio (CD and mp3) formats. Participants will receive a daily email or text reminder to practice the intervention if deemed appropriate. Participants will be given the choice to complete a daily monitoring sheet or have their daily online access monitored to record levels of CFT practice. Participants will be asked to practice the intervention on a daily basis for three weeks with repeated completion of the online assessments and the HRV measurements in the week following the block.

An a priori power calculation was obtained using G*Power 3.1.9 software (Faul, Erdfelder, Buchner & Lang, 2009). With the Depression, Anxiety and Stress Scale (DASS-21: Lovibond & Lovibond, 1995) as the primary outcome measure, the average effect size of a brief CFT intervention on the DASS was equivalent to a large effect size f of .74 (McEwan & Gilbert, 2013). An average estimate of test-retest reliability is 0.77 (Brown, Chorpita, Korotitsch & Barlow, 1997).

Given the number of groups (2) and repetitions (4) in the planned study and assuming a test-retest reliability of .77, a sample size of at least 16 (8 per group) will be required to provide sufficient power (80%) to detect an effect of similar magnitude (f = .74) at an alpha level of .05.

Average attrition rates for clients with PTSD are approximately 20%, although rates vary up to 48% (Imel, Laska, Jakupcak & Simpson, 2013). A cautious 60% (approx.) attrition rate has been considered given the research is additional to participants' involvement at the CTRG. Further allowing room for a more moderate effect size, given that the intervention has not previously been trialled with a clinical sample, a target sample of 40 participants will be sought. Given the 150 referrals received by the CTRG last year this is feasible.

Withdrawal Participants will be assigned a code number with which all of their assessment data will be stored on a password-protected computer file. This will be accessible only to the researcher and any transferring of data will be done using an encrypted memory stick. Any personal data used to contact participants will be deleted upon completion of the experimental aspects of the project. Participants can withdraw at any time but will be informed that any data collected past the first week of the intervention process cannot be erased and may still be used in the project analyses. Consent forms will be signed and will be stored in a locked filing cabinet at the researcher's home office and transferred to the University of Lincoln's archived storage following project completion. Data will be stored for seven years in line with the University's data storage policy.

Implications and Dissemination This research project will contribute to the theoretical literature on both CFT and PTSD. It is anticipated that it will offer new findings regarding self-practice interventions for PTSD which may have beneficial psychological and physiological implications and impact on TAU outcomes. The project will be prepared for publication in an appropriate peer-reviewed journal and presented at relevant conferences. It may also be disseminated on the Compassion Mind Foundation Website.

In the event that any participants find the intervention difficult or experience distress, they will be able to discuss this with an identified person and if deemed appropriate, will be withdrawn from the project. Research suggests continued practice may reduce fear of compassion (Rockliff, et al. 2008) and this information will be shared with participants. It is felt that the risk of such adverse events is minimal.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand verbal and written English language (due to resources, the adapted intervention will not be translated);
* ***To be on the waiting list for therapy at the Centre for Trauma Resilience and Growth, Nottingham UK***;
* Able to access a computer, CD player or mp3 file;
* Had experience of a traumatic event

Exclusion Criteria:

* participants involved in the pilot phase of the project
* unable to understand verbal and written English language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-02; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Depression Anxiety and Stress Scales (DASS-21) | up to six weeks
  21-item version. Self-report measuring negative emotional states of depression, anxiety and stress

SECONDARY OUTCOMES:
Heart Rate Variability (HRV) | three weeks, six weeks
  Measured by the Polar RS800CX Heart Rate Monitor (HRM). This includes the wearing of a watch and chest strap, for which full fitting instructions will be provided to allow participants to complete this procedure with privacy and dignity. Instructions will be reviewed and adapted for the participants if deemed appropriate
Self-Compassion Scale (SCS) | three weeks, six weeks
  A 12-item scale measuring levels of self-compassion
Fears of Compassion Scale (FOC) Scale 3: Expressing kindness and compassion towards yourself. | three weeks, six weeks
  The subscale includes 15 items measuring fears of self-compassion. Permission has been granted by the authors to use in isolation the self-compassion subscale for the research project
The Forms of Self-Criticising/Attacking & Self-Reassuring Scale (FSCRS) | three weeks, six weeks
  22-item self-report questionnaire measuring self-criticism and the ability to self-reassure when things go wrong
Social Safeness and Pleasure Scale (SSPS) | three weeks, six weeks
  The scale measures the extent to which people experience their social worlds as safe, warm and soothing
Impact of Event Scale Revised (IES-R) | up to six weeks
  Evaluates individual's experiences of avoidance and intrusion
Psychological Well-Being - Post-Traumatic Change Questionnaire (PWB-PTCQ) | up to six weeks
  An 18-item self-report questionnaire which assesses participants' perception of changes in psychological well-being after traumatic events

CONTACTS AND LOCATIONS:
Overall Officials: Claire Rycroft, Principal Investigator — University of Lincoln
Locations (1):
- University of Lincoln, Lincoln, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Currently no plans to share IPD. If researchers wish to view data analysis following the study they can contact the researcher.